CLINICAL TRIAL: NCT06528210
Title: Single-Arm, Open-Label, Phase II Study of Pembrolizumab Plus Androgen Deprivation Therapy (ADT) in Combination With Radiotherapy (RT) for High Risk Localized Prostate Cancer
Brief Title: Pembrolizumab With Androgen Deprivation Therapy and Radiotherapy for the Treatment of Patients With High Risk Localized Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Arthur Hung, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025491; NCI-2024-04337 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025491 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-05-30; First posted 2024-07-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: High Risk Prostate Carcinoma; Localized Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Leuprolide; Goserelin; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; relugolix; bicalutamide; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Pembrolizumab, ADT, radiotherapy) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 51 weeks in the absence of disease progression or unacceptable toxicity. Patients receive standard of care ADT with GNRH agonist (leuprolide, goserelin, triptorelin) or GNRH antagonist (relugolix, degarelix) for a total of 24 months, bicalutamide PO QD for 6 months or up to 24 months per the discretion of the treating physician and radiation therapy per standard of care. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo bone scan and/or CT scan/MRI during screening and prostate biopsy and blood sample collection throughout the study.
  Interventions: Drug: Gonadotropin Releasing Hormone Agonists and Antagonists; Drug: Bicalutamide; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: Bone Scan

INTERVENTIONS:
Drug: Gonadotropin Releasing Hormone Agonists and Antagonists — Given PO, IM, Sub-Q injection or Sub-Q implant
  Other Names: GnRH Antagonist; Gonadotropin Releasing Hormone Inhibitor; Leuprolide; Goserelin; Triptorelin; Degarelix; Relugolix
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Procedure: Biopsy Procedure — Undergo prostate biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475
Other: Questionnaire Administration — Ancillary study
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy

SUMMARY:
This phase II trial tests how well pembrolizumab along with standard of care androgen deprivation therapy, with bicalutamide and gonadotropin releasing hormone agonist, and radiotherapy for the treatment of patients with high risk prostate cancer that has not spread to other parts of the body (localized). A monoclonal antibody, such as pembrolizumab, is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Bicalutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of tumor cells. Gonadotropin-releasing hormone agonists prevent the body from making luteinizing hormone-releasing hormone (LHRH) and luteinizing hormone (LH). This causes the testicles to stop making testosterone (a male hormone) in men and may stop the growth of prostate cancer cells that need testosterone to grow. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Giving pembrolizumab with androgen deprivation therapy and radiotherapy may kill more tumor cells in patients with high risk localized prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the rate of prostate biopsy positivity at 6 months (mo.) in patients receiving pembrolizumab plus androgen deprivation therapy (ADT) in combination with radiotherapy.

II. Determine the safety of pembrolizumab in combination with ADT and radiotherapy.

SECONDARY OBJECTIVES:

I. Compare 6-month post-treatment biopsy positive rate in patients stratified by pre-treatment prostate infiltrating T-cell PD-1 and PD-L1 expression.

II. Measures changes in health related quality of life (HRQOL). III. Determine the rate of grade 3 or higher Immune-related adverse events (irAEs).

IV. Determine the rate of biochemical relapse-free survival (bRFS) stratified by tumor PD-1 and PD-L1 expression.

EXPLORATORY OBJECTIVES:

I. Determine the time to cancer-directed treatment in subjects undergoing experimental treatment.

II. Determine the 5-year rate of biochemical relapse-free survival ([bRFS,] i.e. prostate specific antigen [PSA] > nadir + 2 ng/mL) III. Determine the nadir biochemical response rate (nadir PSA ≤ 0.5 ng/mL) IV. Determine the clinical and bRFS at five years. V. Report safety and tolerability of pembrolizumab, defined as pembrolizumab related adverse event of any grade and drug dose modification.

VI. Determine metastases-free survival based on conventional imaging (not positron emission tomography [PET] based).

VII. Determine the serum castration recovery rate (testosterone above 50 ng/dL) VIII. Determine the serum testosterone recovery rate (testosterone above 200 ng/dL) IX. Assess the effect of pembrolizumab combined with ADT + radiation therapy (RT) on serum, blood and tissue markers of the immune response.

X. Correlate changes in markers of inflammatory response with clinical outcomes including post-treatment biopsy rate, PSA response and tumor free survival.

XI. Correlate baseline prostate specific membrane antigen (PSMA) scan findings with efficacy endpoints.

XII. Changes from pre- to post-treatment serum, peripheral blood mononuclear cells (PBMC), blood, microbial and tissue markers of the immune response.

XIII. Correlation of changes in markers of inflammatory response with clinical outcomes including biopsy-complete response, PSA response and disease free survival.

XIV. Determine the rate of local tumor eradication at 12 months for those who had persistent tumor at 6 months.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 51 weeks in the absence of disease progression or unacceptable toxicity. Patients receive standard of care ADT with GNRH agonist (leuprolide, goserelin, triptorelin) or GNRH antagonist (relugolix, degarelix) given orally (PO), subcutaneously (sub-Q) or via sub-Q implant for a total of 24 months, bicalutamide PO once per day (QD) for 6 months or up to 24 months per the discretion of the treating physician and radiation therapy per standard of care. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo bone scan and/or computed tomography (CT) scan/ magnetic resonance imaging (MRI) during screening and prostate biopsy and blood sample collection throughout the study.

After completion of study therapy, patients are followed up at 30 days and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are at least 18 years of age on the day of signing informed consent with newly diagnosed histologically confirmed non-metastatic adenocarcinoma of the prostate (regional spread as defined by National Comprehensive Cancer Network [NCCN] guidelines is allowed) will be enrolled in this study with any one of the following three high risk features:

  * Gleason grade > 8-10
  * PSA > 20 ng/ml
  * Clinical stage T3a or T3b (T4 not allowed, see exclusion criteria)
* Participants must agree to use a contraception as detailed in the protocol during the treatment period and for at least 12 months plus an additional 90 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 30 days prior to the first dose of study intervention
* Absolute neutrophil count (ANC) ≥ 1500/µL. (Specimens must be collected within 10 days prior to the start of study intervention)
* Platelets ≥ 100 000/µL. (Specimens must be collected within 10 days prior to the start of study intervention)
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L. (Specimens must be collected within 10 days prior to the start of study intervention)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine OR measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥ 30 mL/min for participant with creatinine levels > 1.5 × institutional upper limit of normal (ULN). (Specimens must be collected within 10 days prior to the start of study intervention)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin ≤ 1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels > 1.5 × ULN. (Specimens must be collected within 10 days prior to the start of study intervention)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases). (Specimens must be collected within 10 days prior to the start of study intervention)
* International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants. (Specimens must be collected within 10 days prior to the start of study intervention)
* Be willing to undergo a post-treatment prostate biopsy 6 months after completion of therapy on cycle 1 day 1 and optional re-biopsy at 12 months post cycle 1 day 1 if 6-month biopsy was positive for viable tumor
* PSA ≤ 100 ng/mL within 90 days of initiation of therapy. If PSA is repeated and drops below 100 ng/mL without treatment, enrollment will be permitted
* If PSMA PET CT scan shows metastatic spread which is not detected on conventional imaging (CT or bone scan), enrollment is allowed if tumor is considered low volume (≤ 4 sites) with no visceral disease. (PSMA PET CT recommended but not required for enrollment.)
* Must be willing to complete psychosocial and quality of life forms
* Criteria for known hepatitis B and C positive subjects.

  * Hepatitis B and C screening tests are not required unless:

    * Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
    * As mandated by local health authority
* Hepatitis B positive subjects

  * Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
  * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention
* Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

  * Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation
* Has received prior radiotherapy or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-central nervous system (CNS) disease, with a 1-week washout, is permitted
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder that have undergone potentially curative therapy are not excluded
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Concurrent active hepatitis B (defined as HBsAg positive and/or detectable HBV deoxyribonucleic acid [DNA]) and hepatitis C virus (defined as anti-HCV antibody [Ab] positive and detectable HCV ribonucleic acid [RNA]) infection.

Note: Hepatitis B and C screening tests are not required unless:

* Known history of HBV and HCV infection
* As mandated by local health authority

  * Plans to use abiraterone and prednisone in combination with radiotherapy. This must be decided before enrollment
  * Clinical T4 disease is excluded as the primary endpoint cannot be adequately assessed for response in the surrounding tissue based on biopsy
  * Evidence of metastatic, non-regional disease on conventional imaging, including MRI, CT and bone scan
  * Prostate size > 80 cc by MRI or ultrasound
  * Subject has undergone a prior radical prostatectomy. Transurethral resection or other surgical procedure for outlet obstruction allowed
  * Subject has had major surgical procedures within 30 days of allocation
  * Has not adequately recovered from major surgery or has ongoing surgical complications
  * Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
  * Expecting to procreate within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
  * Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Biopsy-complete response determined by post-treatment biopsy | From first dose of pembrolizumab Cycle 1 Day 1 to 6 months after Cycle 1 Day 1. Cycle length is 21 days.
  Will be defined as absence of detectable malignant cells in cores evaluated by established histologic techniques. An exact one-sided confidence interval will also be estimated and provided.
Incidence of adverse events | From first dose of pembrolizumab to 30 days after last dose of pembrolizumab
  Using Common terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Post-treatment cancer detection rates in tumors by levels of PD-1 and PD-L1 expression | From first dose of pembrolizumab to 6 months after Cycle 1 Day 1. Cycle length is 21 days.
  Will be evaluated by pre-treatment prostate infiltrating T-cell PD-1 expression status based on the median split of the expression level. Exact 95% confidence intervals will also be estimated and provided.
Health related quality of life | From screening up to 5 years
  Will be summarized at each appropriate time point using number completed, mean, standard deviation, and 95% confidence intervals.
Incidence of grade 3 or higher immune related adverse events | From first dose of pembrolizumab to 30 days after last dose of pembrolizumab
  Using CTCAE version 5.
Rate of biochemical relapse-free survival | From enrollment of trial to 30 days post last dose of pembrolizumab
  Will be estimated using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Hung, Principal Investigator — OHSU Knight Cancer Institute

IPD SHARING:
Plan to Share IPD: Undecided